CLINICAL TRIAL: NCT05374668
Title: The Effects of Video-based Yoga Interventions on Musculoskeletal Pain and Quality of Life of Patients' Post-corona Virus Disease: a Semi-randomized Controlled Prospective Study
Brief Title: The Effects of Video-based Yoga Interventions for Patients With Post-corona Virus Disease
Acronym: Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Habibe Serap Inal, Prof.Dr., Istinye University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Yoga COVID-19
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Post-COVID-19
Keywords: Pain; Post-COVID-19 patients; Mild symptoms; Quality of life; Functional capacity
MeSH Terms: conditions — Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Semi-randomized controlled prospective study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-based Yoga (Experimental): video-based yoga (n=40) given for patients in post-covid-19 status for 8 weeks
  Interventions: Behavioral: Video-based Yoga Exercises
- Home-based postur exercises (Experimental): Home exzercises were given for 8 weeks
  Interventions: Behavioral: Video-based Yoga Exercises

INTERVENTIONS:
Behavioral: Video-based Yoga Exercises — They were trained face-to-face with social distancing and a maximum of three participants. They were observed while practicing and necessary alerts and corrections were made. Documents related to the videos for yoga exercises and posture exercises specially prepared for this study by the qualified physiotherapist (MD) were provided to the participants
  Other Names: Home-based posture exercises; Control group without any activity

SUMMARY:
Aimed to understand if yoga exercises are superior to posture exercises as an alternative exercise therapy for relieving musculoskeletal pain, improving functional status, and improving quality of life during the post- corona virus disease (COVID-19) period?

DETAILED DESCRIPTION:
Eighty five of 200 post- COVID-19 patients, who met the inclusion/exclusion criteria obtained from the records of the State Hospital. The participants were divided into video-based (VB) yoga (n=40), home-based (HB) posture exercise (n=28), and control (n=17) groups. The socio-demographic characteristics, pain status, walking and balance, and quality of life were evaluated twice, once before and eight weeks after the exercises.

ELIGIBILITY:
Inclusion Criteria:

* recently diagnosed with Covid-19 and discharged from the hospital;
* being at level 0: neglected functional limitation or level 1: negligible functional limitation on the Post-Covid-19 Functional Status Scale,
* referred for physical therapy for musculoskeletal pain.

Exclusion Criteria:

* having any type of surgery in the last six months,
* being pregnant,
* being level 2 or above on the Post-Covid-19 Functional Status Scale

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2022-04-24 (Actual)

PRIMARY OUTCOMES:
Pain Assessment by McGill-Melzack Pain Questionnaire | Baseline
  Assessment of pain by McGill-Melzack Pain Questionnaire: The localization (deep-D; superficial-S) of the pain was determined by a question in the first section of the questionnaire. Subsequently, the features (20 words and 2-6 sub words of each) and severity (mild to unbearable pain, Likert scale-5) of the pain were determined by questions in the second and third section of the questionnaire. In the fourth section, the relationship between pain, time, frequency, and the affecting factors was determined. Scores (total 0-112) obtained from the sections of the survey were collected. The pain level of the patients indicated that the higher the pain, the higher the score.
Balance and gait assessment | At the beginning of the interventions
  Balance and Gait Assessment: The total scores for balance and walking were 0-29 and 0-9, respectively. These scores aimed to reflect the fear of falling. There was no specific cutoff score. As the score increased, the fear of falling decreased.
Quality of life assessment by WHOQOL-BREF | Baseline
  The WHOQOL-short form consists of 26 questions and measures the physical, mental, social, and environmental well-being of the adult population. The Turkish version has 27 questions. The 27th is termed the Environment-Turkish. Each area refers to the quality of life in a respective field independently. The area scores are calculated between 1 and 100 by The World Health Organization Quality of Life-short form: The higher the score, the higher the quality of life.
Muscle Power assessment by handheld dynamometer (MicroFet 2; kgm, Hoggan Scientific, Salt Lake City, UT, USA) | Baseline
  The participants performed maximal isometric voluntary contractions (for lower extremity: M. quadriceps femoris, hamstring group muscles, M. tibialis anterior, M. gastrocnemius, and M. soleus; for upper extremity: M. triceps brachii, M. biceps brachii, and M. deltoideus: anterior, middle, and posterior heads) forcefully against the dynamometer. The dynamometer was held stationary by the physical therapist.
Pain Assessmentby McGill-Melzack Pain Questionnaire | Baseline
  Assessment of pain by McGill-Melzack Pain Questinnaire: The localization (deep-D; superficial-S) of the pain was determined by a question in the first section of the questionnaire. Subsequently, the features (20 words and 2-6 sub words of each) and severity (mild to unbearable pain, Likert scale-5) of the pain were determined by questions in the second and third section of the questionnaire. In the fourth section, the relationship between pain, time, frequency, and the affecting factors was determined. Scores (total 0-112) obtained from the sections of the survey were collected. The pain level of the patients indicated that the higher the pain, the higher the score.
Balance and gait assessment by TBGA | Balance
  Tinetti Balance and Gait Assessment: The total scores for balance and walking were 0-29 and 0-9, respectively. These scores aimed to reflect the fear of falling. There was no specific cutoff score. As the score increased, the fear of falling decreased.
Quality of life assessment of WHOQOL-BREF | Baseline
  The WHOQOL-short form consists of 26 questions and measures the physical, mental, social, and environmental well-being of the adult population. The Turkish version has 27 questions. The 27th is termed the Environment-Turkish. Each area refers to the quality of life in a respective field independently. The area scores are calculated between 1 and 100. by The World Health Organization Quality of Life-short form: The higher the score, the higher the quality of life.
Muscle Power assessment by handheld dynamometer (MicroFet 2; kgm; Hoggan Scientific, Salt Lake City, USA) | Baseline
  The participants performed maximal isometric voluntary contractions (for lower extremity: M. quadriceps femoris, hamstring group muscles, M. tibialis anterior, M. gastrocnemius, and M. soleus; for upper extremity: M. triceps brachii, M. biceps brachii, and M. deltoideus: anterior, middle, and posterior heads) forcefully against the dynamometer. The dynamometer was held stationary by the physical therapist.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Ince DI, Yaglı NV, Saglam M, Kutukcu, EC. Acute and Post-acut Physiotherapy and Rehabilitation in COVI-19 Infection [COVID-19 Enfeksiyonunda Akut ve Post-Akut Fizyoterapi ve Rehabilitasyon]. Turk J Physiother Rehabil. 2020; 31(1):81-93. doi: 10.21653/tjpr.718877.
- [Background] Herrero-Montes M, Fernandez-de-Las-Penas C, Ferrer-Pargada D, Tello-Mena S, Cancela-Cilleruelo I, Rodriguez-Jimenez J, Palacios-Cena D, Paras-Bravo P. Prevalence of Neuropathic Component in Post-COVID Pain Symptoms in Previously Hospitalized COVID-19 Survivors. Int J Clin Pract. 2022 Mar 16;2022:3532917. doi: 10.1155/2022/3532917. eCollection 2022. PMID 35685491
- [Background] Maugeri G, Musumeci G. Adapted Physical Activity to Ensure the Physical and Psychological Well-Being of COVID-19 Patients. J Funct Morphol Kinesiol. 2021 Jan 29;6(1):13. doi: 10.3390/jfmk6010013. PMID 33572883